CLINICAL TRIAL: NCT07319520
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory, Phase II Clinical Trial for the Efficacy Investigation and Safety Evaluation of DW4902 in Patients With Uterine Fibroids
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DW4902
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW4902-201
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myoma of Uterus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo 4 capsules
  Interventions: Drug: DW4902 Placebo
- Low-Dose (Experimental): DW4902 80mg 2 capsules , Placebo 2 capsules
  Interventions: Drug: DW4902 160mg
- Medium-Dose (Experimental): DW4902 80mg 3 capsules , Placebo 1 capsules
  Interventions: Drug: DW4902 240mg
- High-Dose (Experimental): DW4902 80mg 4 capsules
  Interventions: Drug: DW4902 320mg

INTERVENTIONS:
Drug: DW4902 Placebo — Starting from the Baseline Visit (Visit 3), administer orally once daily at a dose of 4 capsules before meals for 12 weeks. (Placebo 4 capsules)
  Arms: Placebo
Drug: DW4902 160mg — Starting from the Baseline Visit (Visit 3), administer orally once daily at a dose of 4 capsules before meals for 12 weeks.. (DW4902 80mg 2 capsules , Placebo 2 capsules)
  Arms: Low-Dose
Drug: DW4902 240mg — Starting from the Baseline Visit (Visit 3), administer orally once daily at a dose of 4 capsules before meals for 12 weeks.. (DW4902 80mg 3 capsules , Placebo 1 capsules)
  Arms: Medium-Dose
Drug: DW4902 320mg — Starting from the Baseline Visit (Visit 3), administer orally once daily at a dose of 4 capsules before meals for 12 weeks.. (DW4902 80mg 4 capsules)
  Arms: High-Dose

SUMMARY:
A Multi-center, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory, Phase II Clinical Trial for the Efficacy Investigation and Safety Evaluation of DW4902 in Patients with Uterine Fibroids.

ELIGIBILITY:
Inclusion Criteria:

- [For Subjects Requiring a Run-in Period]

- Screening Visit 1 (Visit 1) Inclusion Criteria

1. Premenopausal women aged 19 years or older.
2. Subjects diagnosed with uterine fibroids prior to screening, based on imaging studies.
3. At least one uterine fibroid with a longest diameter (D1) ≥3 cm confirmed by transvaginal ultrasound at Screening Visit 1.
4. History or symptoms of heavy menstrual bleeding (HMB) due to uterine fibroids, confirmed prior to screening.
5. Subject agrees to comply with the following contraceptive methods and restrictions during the clinical trial.
6. Subject agrees to use the sanitary products provided during the clinical trial.
7. Subject has voluntarily consented to participate in this clinical trial and signed the informed consent form.

   - Screening Visit 2 (Visit 2) Inclusion Criteria
8. Prior to Screening Visit 2, the subject has had at least two regular menstrual cycles with menstruation lasting at least three consecutive days in each cycle.
9. Subject, in the investigator's clinical judgment, is determined to have symptoms of heavy menstrual bleeding (HMB) due to uterine fibroids, requiring medication.

   * Baseline Visit (Visit 3) Inclusion Criteria
10. During the screening period, the subject has had regular menstrual cycles with menstruation lasting at least three consecutive days in each cycle.
11. During the screening cycle (Pre-C), a PBAC assessment score of 120 or higher is confirmed.

    * [For Subjects Not Requiring a Run-in Period]
    * Screening Visit 2 (Visit 2) Inclusion Criteria

<!-- -->

1. Premenopausal women aged 19 years or older.
2. Subjects diagnosed with uterine fibroids prior to screening via imaging , and at least one uterine fibroid with a longest diameter (D1) ≥3 cm confirmed by transvaginal ultrasound at Screening Visit 2.
3. Subject, in the investigator's clinical judgment, is determined to have symptoms of heavy menstrual bleeding (HMB) due to uterine fibroids, requiring medication.
4. Within 3 months prior to screening, the subject has had regular menstrual cycles with menstruation lasting at least three consecutive days in each cycle.
5. Subject agrees to comply with the following contraceptive methods and restrictions during the clinical trial.
6. Subject agrees to use the sanitary products provided during the clinical trial.
7. Subject has voluntarily consented to participate in this clinical trial and signed the informed consent form.

   - Baseline Visit (Visit 3) Inclusion Criteria
8. During the screening period, the subject has had regular menstrual cycles with menstruation lasting at least three consecutive days in each cycle.
9. During the screening cycle (Pre-C), PBAC assessment score of 120 or higher is assessed.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from participation in this clinical trial.

1. A person who is expected to perform the following surgical (procedure) history during the screening period or during the clinical trial period.

   ① Surgery (procedure) history of uterine fibroids within 24 weeks prior to participation in screening.

   : myomectomy, high intensity focused ultrasound, uterine artery embolization etc.

   ② hysterectomy, ovarian resection, endometrial ablation.

   ③ Surgery that may affect gastrointestinal absorption of clinical trial drugs. However, simple appendectomy and hernia surgery can be participated.
2. As a result of imaging examination at the time of screening (ultrasound, etc.), a person identified as having a gynecological disorder evaluated clinically significant by the examiner other than uterine myoma.
3. During the screening period, the following medical history or comorbidities are identified.

   * Endometriosis or symptomatic dominant adenomyosis.

     * Anovulatory bleeding, non-diagnostic abnormal uterine bleeding, or non-diagnostic abnormal genital bleeding.

       * Lower abdominal pain or pelvic inflammatory disease due to trauma or a condition other than uterine fibroids (e.g., irritable bowel syndrome, interstitial cystitis, etc.) within 12 weeks prior to screening participation.

         * Metabolic bone disease, including osteoporosis.

           * Thyroid/parathyroid disease (e.g., hyperthyroidism, hyperparathyroidism), hyperprolactinemia, anorexia nervosa, which contributes to bone mineral density loss, within 24 weeks prior to screening participation.

             * Any malignancy, including gynecologic cancer, within 5 years prior to screening participation. However, skin basal cell carcinoma/polarized cell carcinoma/microthyroid papillary carcinoma can participate after successful treatment.

               * Type 1 diabetes or uncontrolled type 2 diabetes.

                 * Major cardiovascular disease within 24 weeks prior to screening.

                   * Severe cardiac disease (heart failure (NYHA class 3 and 4), acute coronary artery disease (unstable angina, acute myocardial infarction), clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other arrhythmias deemed clinically significant by the investigator, and peripheral vascular disease.
                   * Hypertrophic obstructive cardiomyopathy, clinically significant valvular heart disease, or aortic disease, etc.

                     * Blood disorders. However, those with iron-deficiency anemia are eligible for participation.

                       * thalassemia, sickle cell anemia, folic acid deficiency, coagulopathy. etc. ⑩ Gastrointestinal diseases that may affect the gastrointestinal absorption of the investigational drug at the time of screening ⑪ Active hepatitis B or active hepatitis C at the time of screening ⑫ History of HIV (human immunodeficiency virus) infection ⑬ History of major psychiatric disorders (such as depression, bipolar disorder), or history of substance/alcohol abuse
4. Subjects exhibiting any of the following test results during the screening period

   * Hemoglobin (Hb) < 8 g/dL (Grade 3 anemia according to CTCAE ver. 5.0)

     * Bone mineral density test (dual energy x-ray absorptiometry, DXA): Z-score ≤ -1.5 in the lumbar spine, total hip, or femoral neck

       * QTc interval > 480 msec* (Grade 2 according to CTCAE ver. 5.0)

         * Fridericia's QT correction formula ④ AST or ALT > 3 x ULN (Grade 2 according to CTCAE ver. 5.0)

           ⑤ Creatinine > 1.5 x ULN (Grade 2 according to CTCAE ver. 5.0)

           ⑥ Uncontrolled hypertension (sitSBP ≥ 160 mmHg or sitDBP ≥ 100 mmHg; Grade 3 according to CTCAE ver. 5.0)

           ⑦ Clinically significant abnormal pathological findings in endometrial biopsy

           ⑧ Positive result from PAP smear test
         * according to Bethesda system >NILM (negative for intraepithelial lesion or malignancy)
5. Pregnant or lactating women during the screening period
6. Subjects with a history of administering or expected to administer the following medications during the clinical trial:

   ① Use of the following medications within 12 weeks prior to Screening Visit 2, or use of hormonal contraceptives within 8 weeks prior to Visit 2(including estrogen/progesterone supplements)/hormonal intrauterine device. However, for medroxy progesterone acetate injection depot formulations and Leuprorelin depot 22.5 mg, 30 mg, or 45 mg, administration within 24 weeks prior to Screening Visit 2 must be confirmed.

   GnRH agonists (e.g., Leuprorelin depot 11.25 mg), GnRH antagonists, selective estrogen receptor modulators, progesterone receptor modulators, anti-gonadotropins, gonadotropin-releasing hormones, aromatase inhibitors, anti-estrogens, prolactin inhibitors, spironolactone, etc. However, administration of Leuprorelin depot 3.75 mg within 4 weeks prior to the screening visit constitutes an exclusion criterion.
   * Use of therapeutic agents for metabolic bone diseases within 12 weeks prior to Screening Visit 2.

     * Use of anticoagulants, antiplatelet agents, or low-dose aspirin within 4 weeks prior to Screening Visit 2

       * Use of antifibrinolytic agents within 4 weeks prior to Screening Visit 2 ⑤ Use of analgesics other than ibuprofen during the clinical trial ⑥ Systemic corticosteroids administered for 14 days or more within 12 weeks prior to Screening Visit 2 ⑦ Strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) within 4 weeks prior to Screening Visit 2 ⑧ Strong inducers or inhibitors of P-glycoprotein (P-gp) within 4 weeks prior to Screening Visit 2
7. Hypersensitivity or allergy to the components of the investigational drug.
8. Hypersensitivity or allergy to hygiene products.
9. Individuals for whom the gynecological examinations required by the study are considered difficult or impossible to perform.
10. Individuals who have participated in other clinical trial and received investigational drugs or investigational medical devices within 4 weeks prior to screening.
11. Individuals otherwise deemed unsuitable for participation in the clinical trial by the investigator.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a total PBAC score | 6 to 12 week period since the baseline visit
  Percentage of subjects with a total PBAC score of less than 10 points in the 6 to 12 week period since the baseline visit

SECONDARY OUTCOMES:
Percentage of subjects with a total PBAC score | 2 to 6 week period since the baseline visit.
  Percentage of subjects with a total PBAC score of less than 10 points in the 2 to 6 week period since the baseline visit.
Percentage of subjects with a total PBAC score | 8 to 12 week period since the baseline visit.
  Percentage of subjects with a total PBAC score of less than 10 points in the 8 to 12 week period since the baseline visit.
Percentage of subjects with a total PBAC score | 12-week visit point after dosing
  Percentage of subjects with a total PBAC score of less than 10 points in the previous recent menstrual cycle, as of the 12-week visit point after dosing
Percentage of subjects for amenorrhea | 6 to 12 week period after the baseline visit
  Percentage of subjects for amenorrhea during the 6 to 12 week period after the baseline visit
Percentage of subjects for amenorrhea | 2 to 6 week period after the baseline visit
  Percentage of subjects for amenorrhea during the 2 to 6 week period after the baseline visit
Changes in hemoglobin levels (g/dL) | 8 weeks and 12 weeks after dosing compared to baseline visits
  Changes in hemoglobin levels (g/dL) at 8 weeks and 12 weeks after dosing compared to baseline visits
The proportion of subjects whose hemoglobin level increased by >2 g/dL | 8 week and 12 week visits compared to the baseline visit
  Among subjects with a hemoglobin level ≤10.5 g/dL at the baseline visit, the proportion of subjects whose hemoglobin level increased by >2 g/dL at the 8-week and 12-week visits compared to the baseline visit
Changes and rates of change in uterine fibroid size | 12 week visit after dosing compared to the baseline visit
  Changes and rates of change in uterine fibroid size at the 12-week visit after dosing compared to the baseline visit
Changes and rates of change in uterine size | 12 week visit after dosing compared to the baseline visit
  Changes and rates of change in uterine size at the 12-week visit after dosing compared to the baseline visit
The proportion of subjects with a uterine fibroid-associated peak NRS pain score | 6 to 12 week period after the baseline visit
  Among subjects with a uterine fibroid-associated peak NRS pain score of ≥4 during the menstrual cycle (Pre-C) of the screening period, the proportion of subjects with a uterine fibroid-associated peak NRS pain score of ≤1 during the 6 to 12 week period after the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Sunghoon Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No